CLINICAL TRIAL: NCT06279637
Title: Joint Patient and Caregiver Intervention for Older African Americans With Poorly Controlled Type 2 Diabetes (Joint Home-DM-BAT)
Brief Title: Joint Patient and Caregiver Intervention for Older African Americans With Type 2 Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Aprill Z. Dawson, PhD, MPH, Associate Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: PRO00046457
Record Dates: First submitted 2024-02-19; First posted 2024-02-28 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Joint Home-DM-BAT Intervention (Experimental): A trained health educator will deliver the manualized Joint Home-DM-BAT intervention. Participants will receive 8-weekly sessions of diabetes education, problem solving around social needs, and behavioral activation via telephone; and 3 monthly booster sessions.
  Interventions: Behavioral: Joint Home-DM-BAT Intervention
- Usual Care (Active Comparator): Patients randomized to the usual care arm will receive weekly mailings of diabetes education modules for 8 weeks and monthly mailings for 3 months to match the weekly and monthly booster sessions.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Joint Home-DM-BAT Intervention — 8 weekly sessions of telephone-delivered, manualized education on diabetes management, problem solving of social needs, and behavioral activation.
  Arms: Joint Home-DM-BAT Intervention
Behavioral: Usual Care — Diabetes education materials will be mailed weekly and monthly according to the booster schedule
  Arms: Usual Care

SUMMARY:
This study will test the preliminary efficacy of a joint patient/informal caregiver telephone-delivered intervention that includes diabetes education; problem solving around social needs; and behavioral activation for older African Americans with poorly controlled type 2 diabetes by randomizing 100 patient/caregiver dyads to the Joint Home intervention (n=50) and usual care (n=50) arms.

The aims of the study are:

Aim 1: To test the preliminary efficacy of home-based, joint patient and caregiver intervention (Joint Home-DM-BAT) on patient clinical outcomes (hemoglobin A1c, blood pressure, and LDL-Cholesterol).

Aim 2: To test the preliminary efficacy of home-based, joint patient and caregiver intervention (Joint Home-DM-BAT) Joint Home DM-BAT on patient quality of life.

Aim 3: To test the preliminary efficacy of home-based, joint patient and caregiver intervention (Joint Home-DM-BAT) on caregiver quality of life and caregiver burden.

ELIGIBILITY:
Patient Inclusion Criteria:

1. Age ≥50 years of age;
2. Self-identified as Black/African American;
3. Clinical diagnosis of T2DM and poorly controlled, defined as HbA1c ≥8% at the screening visit;
4. Able to communicate in English; and
5. Has an informal caregiver (family member or close friend willing to participate in the study for 6 months.

Caregiver Inclusion Criteria:

1. Willing to attend 4, one-hour sessions with the study participant;
2. Willing to support the study participant for study duration (6 months); and
3. Willing to complete brief baseline, 3- and 6-month assessments.

Patient/Caregiver Exclusion Criteria:

1. Mental confusion at screening assessment suggesting significant dementia;
2. Alcohol or drug abuse/dependency at screening assessment;
3. Active psychosis or acute mental disorder at screening assessment; and
4. Life expectancy <6 months at screening.

Ages: 50 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Glycemic Control (Hemoglobin A1C [HbA1C]) | Change in baseline HbA1C at 6 months post intervention follow-up
  About 10cc of blood will be drawn by trained phlebotomists and sent to the lab for testing.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No